CLINICAL TRIAL: NCT02611882
Title: Evaluation of Gallium-68 HBED-CC-PSMA Imaging in Prostate Cancer Patients
Brief Title: Evaluation of Gallium-68-HBED-CC-PSMA Imaging in Prostate Cancer Patients
Acronym: PSMA PET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Principal Investigator, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 15554; NCI-2018-00037 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2015-09-29; First posted 2015-11-23 (Estimated); Results first posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-11

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — gallium 68 PSMA-11; Positron-Emission Tomography; Tomography, X-Ray Computed; Positron Emission Tomography Computed Tomography; Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- High-risk prostate cancer pre-prostatectomy (preRP) population (Experimental): Patients with high-risk prostate cancer pre-prostatectomy.
  Patients receive Ga-68-HBED-CC-PSMA and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Interventions: Drug: Ga-68 labeled HBED-CC PSMA; Device: Positron Emission Tomography (PET) image combined with Computed Tomography (CT) (PET/CT); Device: Positron Emission Tomography (PET) image combined with Magnetic Resonance Imaging (MRI) (PET/MRI)
- Biochemical Recurrence (BCR) (Experimental): Patients with prostate cancer with biochemical recurrence
  Patients receive Ga-68-HBED-CC-PSMA and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Interventions: Drug: Ga-68 labeled HBED-CC PSMA; Device: Positron Emission Tomography (PET) image combined with Computed Tomography (CT) (PET/CT); Device: Positron Emission Tomography (PET) image combined with Magnetic Resonance Imaging (MRI) (PET/MRI)
- Castrate Resistant Prostate cancer (CRCP) population (Experimental): Patients with castrate resistant prostate cancer.
  Patients receive Ga-68-HBED-CC-PSMA and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
  Interventions: Drug: Ga-68 labeled HBED-CC PSMA; Device: Positron Emission Tomography (PET) image combined with Computed Tomography (CT) (PET/CT); Device: Positron Emission Tomography (PET) image combined with Magnetic Resonance Imaging (MRI) (PET/MRI)

INTERVENTIONS:
Drug: Ga-68 labeled HBED-CC PSMA — The imaging agent (Ga-68 HBED-CC PSMA) will be administered on an outpatient basis. It will be administered a single time intravenously prior to the PET/CT imaging. The one-time nominal injected dose will be 3 to 7 millicurie (mCi) containing 10 - 25 μg Ga-68 HBED-CC PSMA.
  Other Names: Ga-68 labeled DKFZ-PSMA-11; Ga-68 labeled Glu-NH-CO-NH-Lys(Ahx)-HBED-CC; Ga-68 labeled Glu-urea-Lys(Ahx)-HBED-CC
Device: Positron Emission Tomography (PET) image combined with Computed Tomography (CT) (PET/CT) — Patient shall begin imaging between 55 and 70 minutes after the injection of the radiopharmaceutical. A PET/CT scan includes two parts: a PET scan and a CT scan. The CT portion of the scan produces a 3-D image that shows a patient's anatomy. The PET scan demonstrates function and what's occurring on a cellular level. The PET scan is unique because it images the radiation emitted from the patient while the CT records anatomical x-rays, showing the same area from another perspective
  Other Names: PET/CT
Device: Positron Emission Tomography (PET) image combined with Magnetic Resonance Imaging (MRI) (PET/MRI) — Patient shall begin imaging between 55 and 70 minutes after the injection of the radiopharmaceutical. A PET/MRI scan is a two-in-one test that combines images from a positron emission tomography (PET) scan and a magnetic resonance imaging (MRI) scan. Coverage for the scan will extend from the patients vertex through the mid thighs. We will use 4 minute acquisitions per bed position for PET imaging.
  Other Names: PET/MRI

SUMMARY:
The investigators are imaging patients with prostate cancer using a new PET imaging agent (Ga-68 HBED-CC PSMA) in order to evaluate it's ability to detection prostate cancer in patients with high risk disease prior to prostatectomy, patients with biochemical recurrence and patients with castrate resistant prostate cancer.

DETAILED DESCRIPTION:
Imaging and staging of prostate cancer is critical for surgical and treatment planning. Patients with suspected metastatic prostate cancer will be imaged using Gallium-68 labeled HBED-CC PSMA in order to demonstrate its utility. The investigators plan to utilize this data to obtain further approvals of the HBED-CC PSMA compound, so that this agent will become available for clinical imaging in prostate cancer patients.

This compound has been shown to be superior to choline based PET agents for the staging of prostate cancer, both Carbon-11 and Fluorine-18 compounds. But this compound was not patented and therefore no company or private entity will make the investment required to bring HBED-CC PSMA to market. In the vacuum of availability, academic groups must take the lead in order to collect the necessary data for future FDA approval.

This study focuses on three patients populations that are imaged. In the pre-prostatectomy population, the primary objective is to determine the sensitivity and specificity for detection on nodal metastasis. In the biochemical recurrence population, the primary objective is to determine the sensitivity of recurrence location. In the castrate resistant prostate cancer population the primary objective is to determine if PSMA PET detects more metastatic lesions than conventional imaging.

ELIGIBILITY:
Inclusion Criteria:

1. Known prostate cancer with a clinical concern for the presence of metastatic disease as delineated below:

   * Treatment naïve patients with one of the following risk factors: CAPRA (Cancer of the Prostate Risk Assessment) score ≥ 5, Prostate-specific antigen (PSA) ≥ 15 ng/mL and/or Gleason score ≥ 4+4.
   * Patients with biochemical recurrence after prostatectomy or radiation therapy with a PSA doubling time less than 12 months.

     i. These patients may have received androgen deprivation therapy prior to imaging.
   * Patients with castrate resistant prostate cancer with progressive disease as defined by Prostate Cancer Clinical Trials Working Group (PCWG2) criteria (27).

     i. Patients with castrate resistant prostate cancer can be either on treatment or off treatment
2. Age > 18.
3. Karnofsky performance status of > 50 (or Eastern Cooperative Oncology Group (ECOG)/World Health Organization (WHO) equivalent).
4. Ability to understand a written informed consent document, and the willingness to sign it.

Exclusion Criteria:

1. Patients exceeding the weight limitations of the scanner or are not able to enter the bore of the PET scanner due to BMI.
2. Inability to lie still for the entire imaging time (e.g. cough, severe arthritis, etc.).
3. Inability to complete the needed investigational due to other reasons (severe claustrophobia, radiation phobia, etc.).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2015-12-18 (Actual); Primary Completion 2016-10-24 (Actual); Study Completion 2016-10-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hope, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lawhn-Heath C, Flavell RR, Behr SC, Yohannan T, Greene KL, Feng F, Carroll PR, Hope TA. Single-Center Prospective Evaluation of 68Ga-PSMA-11 PET in Biochemical Recurrence of Prostate Cancer. AJR Am J Roentgenol. 2019 Aug;213(2):266-274. doi: 10.2214/AJR.18.20699. Epub 2019 Apr 30. PMID 31039025
- [Derived] Djaileb L, Armstrong WR, Thompson D, Gafita A, Farolfi A, Rajagopal A, Grogan TR, Nguyen K, Benz MR, Hotta M, Barbato F, Ceci F, Schwarzenbock SM, Unterrainer M, Zacho HD, Juarez R, Cooperberg M, Carroll P, Washington S, Reiter RE, Eiber M, Herrmann K, Fendler WP, Czernin J, Hope TA, Calais J. Presurgical 68Ga-PSMA-11 Positron Emission Tomography for Biochemical Recurrence Risk Assessment: A Follow-up Analysis of a Multicenter Prospective Phase 3 Imaging Trial. Eur Urol. 2023 Dec;84(6):588-596. doi: 10.1016/j.eururo.2023.06.022. Epub 2023 Jul 21. PMID 37482512
- [Derived] Hope TA, Eiber M, Armstrong WR, Juarez R, Murthy V, Lawhn-Heath C, Behr SC, Zhang L, Barbato F, Ceci F, Farolfi A, Schwarzenbock SM, Unterrainer M, Zacho HD, Nguyen HG, Cooperberg MR, Carroll PR, Reiter RE, Holden S, Herrmann K, Zhu S, Fendler WP, Czernin J, Calais J. Diagnostic Accuracy of 68Ga-PSMA-11 PET for Pelvic Nodal Metastasis Detection Prior to Radical Prostatectomy and Pelvic Lymph Node Dissection: A Multicenter Prospective Phase 3 Imaging Trial. JAMA Oncol. 2021 Nov 1;7(11):1635-1642. doi: 10.1001/jamaoncol.2021.3771. PMID 34529005
- [Derived] Hope TA, Aggarwal R, Chee B, Tao D, Greene KL, Cooperberg MR, Feng F, Chang A, Ryan CJ, Small EJ, Carroll PR. Impact of 68Ga-PSMA-11 PET on Management in Patients with Biochemically Recurrent Prostate Cancer. J Nucl Med. 2017 Dec;58(12):1956-1961. doi: 10.2967/jnumed.117.192476. Epub 2017 May 18. PMID 28522741

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through clinicians located at San Francisco Veteran's Affairs Medical Center and University of California, San Francisco Helen Diller Family Comprehensive Cancer Center
Groups:
- Biochemical Recurrence (BCR) Population: Patients with prostate cancer with biochemical recurrence.
  Patients receive Ga-68-HBED-CC-PSMA and then undergo PET/CT or PET/MRI approximately 55-70 minutes later.
Period: Overall Study
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population | Castrate Resistant Prostate Cancer (CRCP) Population
Started | 75 | 150 | 0
Completed Surgery Per Protocol (Applies only to participants in the preRP group) | 42 | 0 | 0
Completed | 42 | 150 | 0
Not Completed | 33 | 0 | 0
Not completed — Did not complete prostatectomy per protocol stipulation | 33 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No participants were enrolled in the CRCP arm of this protocol
Groups:
- Total: Total of all reporting groups
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population | Castrate Resistant Prostate Cancer (CRCP) Population | Total
Number analyzed (Participants) | 75 | 150 | 0 | 225
Age, Customized [Count of Participants; unit: Participants]
  40-49 years old | 1 | 1 |  | 2
  50-59 years old | 15 | 14 |  | 29
  60-69 years old | 28 | 60 |  | 88
  70-79 years old | 29 | 64 |  | 93
  80-89 years old | 2 | 10 |  | 12
  90-99 years old | 0 | 1 |  | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 |  | 0
  Male | 75 | 150 |  | 225
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 4 |  | 73
  Not Hispanic or Latino | 2 | 130 |  | 132
  Unknown or Not Reported | 4 | 16 |  | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 61 | 0 |  | 61
  Asian | 3 | 5 |  | 8
  Native Hawaiian or Other Pacific Islander | 1 | 1 |  | 2
  Black or African American | 0 | 1 |  | 1
  White | 0 | 125 |  | 125
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 10 | 18 |  | 28
Region of Enrollment [Number; unit: participants]
  United States | 75 | 150 |  | 225

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of Ga-68 HBED-CC PSMA for Detection of Nodal Metastases
Description: Patients who have a positive node on imaging and on pathology will be considered a true-positive. Patients who have no nodes on imaging and pathology will be considered true- negatives. Patients with positive nodes on imaging and negative on pathology will be considered false positives and those with positive nodes on pathology but negative on imaging will be considered false negatives. Point estimate of the true positive rate will be calculated with the corresponding 95% confidence interval.
Time Frame: 1 day
Measure: Number; unit: proportion of participants
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population
Number analyzed (Participants) | 42 | 72
proportion of participants | .59 | .89

2. Primary Outcome: Specificity of Ga-68 HBED-CC PSMA for Detection of Nodal Metastasis
Description: Patients who have a positive node on imaging and on pathology will be considered a true-positive. Patients who have no nodes on imaging and pathology will be considered true- negatives. Patients with positive nodes on imaging and negative on pathology will be considered false positives and those with positive nodes on pathology but negative on imaging will be considered false negatives. Point estimate of the true negative rate will be calculated with the corresponding 95% confidence interval.
Time Frame: 1 day
Measure: Number; unit: proportion of participants
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population
Number analyzed (Participants) | 42 | 72
proportion of participants | .80 | .31

3. Primary Outcome: Positive Predictive Value (PPV) of Ga-68 HBED-CC PSMA for Detection of Nodal Metastasis
Description: as for outcome 2
Time Frame: 1 day
Measure: Number; unit: proportion of true positives
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population
Number analyzed (Participants) | 42 | 72
proportion of true positives | .67 | .906

4. Primary Outcome: Negative Predictive Value (NPV) of Ga-68 HBED-CC PSMA for Detection of Nodal Metastasis
Description: as for outcome 2
Time Frame: one month
Measure: Number; unit: proportion of true negatives
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population
Number analyzed (Participants) | 42 | 77
proportion of true negatives | .74 | .24

5. Secondary Outcome: Overall Detection Rates of Ga68-PSMA-11 by PSA Levels for the BCR Group
Description: 68Ga-labeled prostate-specific membrane antigen 11 (Ga68-PSMA-11) PET positivity rate by prostate-specific antigen (PSA) level is calculated by the number of positive reads divided by the total number of patients in the BCR Group per PSA value quintile (Detection rate (d) = total number of positive reads (t)/ total number of participants (N)).
Time Frame: Up to 1 year
Population: Six patients did not have an evaluable PSA value pre-imaging for this analysis
Measure: Number; unit: proportion of participants
Arm/Group | Biochemical Recurrence (BCR) Population
Number analyzed (Participants) | 144
proportion of participants
  <0.5 ng/dl | .55
  0.5 to < 1.0 ng/dl | .62
  1.0 to < 2.0 ng/dl | .80
  2.0 to < 5.0 ng/dl | .88
  >=5.0 ng/dl | .96

6. Secondary Outcome: Number of Patients in Biochemical Recurrence (BCR) Group Who Had a Reported Change in Medical Management
Description: Change in participant medical management was determined based on the results of surveys given to each participant's treating physician. Results of the survey were categorized as a major change in participant's medical management, a minor change in participant's medical management, no change to participant's medical management, or change to participant's medical management is unknown. These categories were developed based on a predetermined categorization schema.
Time Frame: Up to 1 year
Population: Surveys for only 126 BCR participants were completed by their physicians
Measure: Count of Participants; unit: Participants
Arm/Group | Biochemical Recurrence (BCR) Population
Number analyzed (Participants) | 126
Participants
  Major Change | 67
  Minor Change | 8

ADVERSE EVENTS:
Time Frame: Up to one year
Arm/Group | High-risk Prostate Cancer Pre-prostatectomy (preRP) Population | Biochemical Recurrence (BCR) Population
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/150
Serious Adverse Events (participants affected / at risk) | 0/75 | 0/150
Other Adverse Events (participants affected / at risk) | 0/75 | 0/150

LIMITATIONS AND CAVEATS:
Over one-half of the patients subsequently underwent radiation therapy and androgen deprivation therapy. In these patients PSA level almost universally falls to zero, and therefore no follow-up imaging is performed, effectively removing a large proportion of patients from our imaging follow-up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes